CLINICAL TRIAL: NCT02167958
Title: Nonmyeloablative Hematopoietic Cell Transplantation (HCT) for Patients With Hematologic Malignancies Using Related, HLA-Haploidentical Donors: A Pilot Trial of Peripheral Blood Stem Cells (PBSC) as the Donor Source
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rafic Farah, MD (Other)
Responsible Party: Sponsor-Investigator, Rafic Farah, MD, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-131
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Leukemia; MDS; Myelofibrosis; Lymphoma
MeSH Terms: conditions — Leukemia; Primary Myelofibrosis; Lymphoma | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Mesna; Whole-Body Irradiation; Stem Cell Transplantation; Tacrolimus; Mycophenolic Acid; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Day -6, -5 Fludarabine 30 mg/M2 IV over 30-60 minutes Cyclophosphamide 14.5 mg/kg IV over 1-2 hours*, Mesna 14.5 mg/kg IV in 4 divided doses
  Day -4 through -2 Fludarabine 30 mg/M2 IV over 30-60 minutes
  Day -1 Total Body Irradiation 200 cGy, donor apheresis
  Day 0 T cell replete PBSC
  Days 3, 4 Cyclophosphamide 50 mg/kg IV Mesna 50 mg/kg IV in 4 divided doses
  Day 5 Begin tacrolimus ,mycophenolate, and G-CSF
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mesna; Radiation: Total Body Irradiation; Other: Hematopoietic stem cell infusion; Drug: Tacrolimus; Drug: Mycophenolate; Drug: G-CSF

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 30 mg/m2/day will be administered over 30-60 minutes intravenous infusion on Days -6 through -2. Fludarabine will be dosed according to the recipient's Adjusted Ideal Body Weight (AIBW) unless AIBW is less than Ideal Body Weight (IBW).
  For decreased creatinine clearance (< 61 mL/min) determined by the Cockcroft Formula:
  Cockcroft-Gault CrCl = (140-age) * (Wt in kg) * (0.85 if female) / (72 * Cr)
  Fludarabine dosage should be reduced per standard of care.
  Other Names: Fludara
Drug: Cyclophosphamide — Pre-transplant
  Cy 14.5 mg/kg/day will be administered as a 1-2 hour intravenous infusion with a high volume fluid flush on Days -6 and -5. Cy will be dosed according to the recipient's actual body weight unless the patient weighs more than 125% of IBW, in which case the drug will be dosed according to the adjusted IBW
  Post-transplant
  Hydration prior to cyclophosphamide may be given according to Standard Practice Guidelines.
  Cyclophosphamide [50mg/kg] will be given on Day 3 post-transplant (between 60 and 72 hours after marrow infusion) and on Day 4 post-transplant (approximately 24 hours after Day 3 cyclophosphamide). Cy will be dosed according to the recipient's actual body weight unless the patient weighs more than 125% of IBW, in which case the drug will be dosed according to the adjusted IBW. Cyclophosphamide will be given as an IV infusion over 1-2 hours.
  .
Drug: Mesna — Pre-transplant
  Mesna should be given in divided doses IV 30 min pre- and at 3, 6, and 8 hours post-cyclophosphamide. Mesna dose will be based on the cyclophosphamide dose being given. The total daily dose of mesna is equal to 100% of the total daily dose of cyclophosphamide.
  Post-transplant
  Mesna should be given in divided doses IV 30 min pre- and at 3, 6, and 8 hours post-cyclophosphamide. Mesna dose will be based on the cyclophosphamide dose being given. The total daily dose of mesna is equal to 100% of the total daily dose of cyclophosphamide.
  Other Names: Mesnex
Radiation: Total Body Irradiation — 200 cGy will be administered in a single fraction on Day -1 via linear accelerator.
Other: Hematopoietic stem cell infusion — Donors who consent to PBSC donation will receive 5 daily doses of G-CSF, 10 μg/kg/day by subcutaneous injection commencing on day -5. PBSC's will be collected in the afternoon of day -1, stored at 4C overnight, and infused as soon as possible on day 0. If the collection on day -1 contains less than 5.0 X 106 CD34+ cells per kg recipient weight, a second collection will be performed the following morning and infused on day 0. Quantitation of CD34 and CD3 cells will be performed by the Cellular Therapy Lab. For all patients, the target number of CD34 cells to be infused should be 5-6 X 106 cells per kg recipient weight. PBSC in excess of 6.0 x 106 CD34 cells/kg recipient weight may be cryopreserved.
  Other Names: PBSC
Drug: Tacrolimus — Tacrolimus will be given at a dose of .03 mg/kg IV over 24 hours. Tacrolimus will be changed to a PO dosing schedule once a therapeutic level is achieved and the patient is tolerating PO. Whole bloodblood levels of tacrolimus will be measured around Day 7 and then should be checked at least weekly thereafter and the dose adjusted accordingly to maintain a level of 5-10 ng/mL. Tacrolimus will be discontinued after the last dose around Day 180, or may be continued if active GVHD is present. Cyclosporine (target concentration 200-400 ng/ml) may be substituted for tacrolimus if the patient is intolerant of tacrolimus.
  Other Names: Astagraf XL; Hecoria; Prograf
Drug: Mycophenolate — Either the sodium salt of mycophenolate or mycophenolate mofetil (MMF) may be used as prophylaxis of GvHD and will be dosed by actual bodyweight. Only MMF is available as IV formulation. Sodium mycophenolate will be given at a dose of 10mg/kg PO TID rounded to the nearest number of 180mg tablets. MMF will be given at a dose of 15 mg/kg PO TID. The maximum total daily dose should not exceed 2160 mg (sodium salt) or 3 grams (mofetil). Mycophenolate prophylaxis will be discontinued after the last dose on Day 35, or may be continued if active GVHD is present.
  Other Names: CellCept; Myfortic
Drug: G-CSF — G-CSF will be given beginning on Day 5 at a dose of 5 mcg/kg/day (rounding to the nearest vial dose is allowed), until the absolute neutrophil count (ANC) is > 1,000/mm3 for three consecutive days.
  Other Names: Granulocyte - Colony Stimulating Factor; Filgrastim; Neupogen®

SUMMARY:
The purpose of this study is to determine whether stem cells collected from a donor's blood stream will be as safe and effective as using bone marrow collected from a donor's pelvic bone.

DETAILED DESCRIPTION:
This is a pilot study to assess the safety and potential efficacy of haploidentical peripheral blood stem cell transplantation using a nonmyeloablative preparative regimen and post-transplant cyclophosphamide. The overall objective of this study is to collect the efficacy and safety data to provide the basis to decide whether a larger study of clinical efficacy is warranted in this setting.

ELIGIBILITY:
Inclusion Criteria:

Subject

1. Age< 70.
2. Molecular based HLA typing will be performed for the HLA-A, -B, -Cw, DRB1 and -DQB1 loci to the resolution adequate to establish haplo identity. A minimum match of 5/10 is required. An unrelated donor search is not required for a patient to be eligible for this protocol if the clinical situation dictates an urgent transplant. Clinical urgency is defined as 6-8 weeks from referral or low-likelihood of finding a matched, unrelated donor.
3. Subjects must meet one of the disease classifications listed below:

   Acute leukemias (includes T lymphoblastic lymphoma). Remission is defined as < 5% blasts with no morphological characteristics of acute leukemia (e.g., Auer Rods) in a bone marrow with > 20% cellularity, peripheral blood counts showing ANC >1000/ul, including patients in CRp.

   Acute Lymphoblastic Leukemia in high risk CR1 as defined by at least one of the following:

   Adverse cytogenetics such as t(9;22), t(1;19), t(4;11), MLL rearrangements White blood cell counts >30,000/mcL Patients over 30 years of age Time to complete remission >4 weeks Presence of extramedullary disease

   Acute Myelogeneous Leukemia in high risk CR1 as defined by at least one of the following:

   Greater than 1 cycle of induction therapy required to achieve remission Preceding myelodysplastic syndrome (MDS) Presence of Flt3 abnormalities FAB M6 or M7 leukemia or

   Adverse cytogenetics for overall survival such as:

   those associated with MDS Complex karyotype (≥ 3 abnormalities) Any of the following: inv(3) or t(3;3), t(6;9), t(6;11), + 8 [alone or with other abnormalities except for t(8;21), t(9;11), inv(16) or t(16;16)], t(11;19)(q23;p13.1)

   Acute Leukemias in 2nd or subsequent remission

   Biphenotypic/Undifferentiated Leukemias in 1st or subsequent CR.

   High-risk MDS status-post cytotoxic chemotherapy

   Myelofibrosis

   Burkitt's lymphoma: second or subsequent CR.

   Lymphoma.

   Chemotherapy-sensitive (complete or partial response; see response criteria Appendix C) large cell, Mantle Cell or Hodgkin's lymphomas that have failed at least 1 prior regimen of multi-agent chemotherapy and are ineligible for an autologous transplant or relapsed/progressed after autologous stem cell transplant.

   Marginal zone B-cell lymphoma or follicular lymphoma that has progressed after at least two prior therapies (excluding single agent Rituxan) and are ineligible for an autologous transplant or relapsed/progressed after autologous stem cell transplant..
4. Patients with adequate physical function as measured by:

   Cardiac: left ventricular ejection fraction at rest must be ≥ 35%.

   Hepatic: bilirubin ≤ 2.5 mg/dL; and ALT, AST, and Alkaline Phosphatase < 5 x ULN.

   Renal: serum creatinine within normal range for age, or if serum creatinine outside normal range for age, then renal function(creatinine clearance or GFR) > 40 mL/min/1.73m2.

   Pulmonary: FEV1, FVC, DLCO (diffusion capacity) ≥ 40% predicted (corrected for hemoglobin); if unable to perform pulmonary function tests, then O2 saturation > 92% on room air.

   Performance status: Karnofsky/Lansky score ≥ 60%.
5. Patients who have received a prior allogeneic HSCT and who have either rejected their grafts or who have become tolerant of their grafts with no active GVHD requiring immunosuppressive therapy.

Donor

1. Donors must be HLA-haploidentical first-degree or second degree relatives of the patient.
2. Age ≥ 18 years
3. Weight ≥ 40 kg

Exclusion Criteria:

Subject

1. HLA-matched donor able to donate.
2. Pregnancy or breast-feeding.
3. Current uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiologic findings).

Donor

1) Positive anti-donor HLA antibody.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2019-09-21 (Actual); Study Completion 2019-09-21 (Actual)

PRIMARY OUTCOMES:
Acute GvHD | Day +84
  The cumulative incidence of grades III/IV acute GvHD at day +84 will be assessed. The first day of acute GvHD onset will be used to calculate a cumulative incidence curve by certain grade. An overall cumulative incidence curve will be computed along with a 90% CI with graft failure, relapse/progression, and death as competing risks.
Chronic Graft-versus-Host Disease | 1 year
  The cumulative incidence of chronic GvHD at one year will be assessed. An overall cumulative incidence curve will be computed along with a 90% CI with graft failure, relapse/progression, and death as competing risks.
Nonrelapse Mortality (NRM) | 1 year
  The cumulative incidence of NRM at 1 year will be assessed. An overall cumulative incidence curve will be computed along with a 90% CI with relapse/progression as competing risk.
Relapse of Malignancy | 1 year
  The cumulative incidence of relapse at 1 year will be assessed. An overall cumulative incidence curve will be computed along with a 90% CI with NRM as competing risk.

SECONDARY OUTCOMES:
Neutrophil Recovery | Up to day +84
  Achievement of an ANC ≥ 500/mm3 for three consecutive measurements on different days. The first of the three days will be designated the day of neutrophil recovery.
Primary graft failure | Day +84
  Primary graft failure < 5% donor CD3 chimerism
Secondary graft failure | Up to 1 year
  Initial recovery followed by neutropenia with < 5% donor chimerism.
Platelet recovery | Up to day +84
  The first day of a sustained platelet count >20,000/mm3 with no platelet transfusions in the preceding seven days.
Donor Cell Engraftment | Day +28, Day >= +84
  Donor chimerism >= 50% on day >= 84 after transplantation. Donor engraftment also should be tested on day +28.
Progression-free Survival | Up to 1 year
  Progression-free survival is the minimum time interval to relapse/recurrence, to death or to last follow-up.
Infections | Date of onset
  Infections will be reported by anatomic site, date of onset, organism and resolution, if any.

CONTACTS AND LOCATIONS:
Overall Officials: Rafic J Farah, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States